CLINICAL TRIAL: NCT00957502
Title: A Prospective, Limited-Use Evaluation of the ENTact™ Septal Stapler for Tissue Approximation Utilizing Staples With Extended Shelf Life
Brief Title: ENTact™ Septal Stapler Shelf Life Extension
Acronym: SSLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ENTrigue Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSA2009-03
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Deviated Nasal Septum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One year aged staples (Experimental): Subjects implanted with sterile staples aged to approximately one year.
  Interventions: Device: ENTact™ Septal Stapler
- 18 month aged staples (Experimental): Subjects implanted with sterile staples aged to approximately 18 months.
  Interventions: Device: ENTact™ Septal Stapler

INTERVENTIONS:
Device: ENTact™ Septal Stapler — 1 year aged septal staples
  Arms: One year aged staples
Device: ENTact™ Septal Stapler — 18 Month Aged Staples
  Arms: 18 month aged staples

SUMMARY:
This study is a prospective, limited-use evaluation of the ENTact™ Septal Stapler for tissue approximation utilizing staples with extended shelf life. The ENTact™ Septal Stapler will be used to approximate the mucoperichondrial flaps in all patients. Each treatment group will be implanted with product that has been aged for a specified amount of time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, between the ages of 18 and 65 years, with a clinically significant deviation of the nasal septum.
* Patient is able to provide a signed informed consent form.
* Patient will agree to comply with all study related procedures.
* Subject is not pregnant at this time by confirmation of one of the following:

  * subject is male,
  * subject not of child bearing age,
  * subject is surgically sterile,
  * subject is not pregnant per negative hCG test.
* Subject does not plan on becoming pregnant and is not breast feeding during the course of the study.

Exclusion Criteria:

* Patients who have had previous septoplasty
* Patients with uncontrolled diabetes
* Presence of infection at the study site
* Subject is a:

  * smoker,
  * severe drug abuser,
  * severe alcohol abuser.
* Patient with autoimmune disease deemed clinically significant by the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Clinical performance of aged ENTact™ Septal Staples | One week post op

SECONDARY OUTCOMES:
Clinical evaluation of gross tissue appearance at implantation site(s) | One week post op
ENTact™ Septal Staple functionality based on maintained coaptation | One week post op

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Tami, MD, Principal Investigator — Good Samaritan Hospital
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States